CLINICAL TRIAL: NCT03066050
Title: Long-Term Follow-Up For Participants Of: Evaluation Of Outcomes Following Mitral Valve Repair/Replacement In SMR and Surgical Interventions For MMR Trials
Brief Title: Long Term Follow Up for CTSN Mitral Valve Repair Studies
Status: Active, not recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Annetine Gelijns, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 08-1078-00012; U01HL088942 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Mitral Valve Insufficiency; Coronary Artery Disease
Keywords: Ischemic Mitral Regurgitation; Mitral Valve Disease; Moderate Mitral Regurgitation; Severe Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Coronary Artery Disease | interventions — Mitral Valve Annuloplasty; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SMR MV Repair: This group of patients had been randomized in the SMR study to mitral valve repair with annuloplasty ring.
  Interventions: Other: MV Repair
- MV Replacement: This group of patients had been randomized in the SMR study to mitral valve replacement.
  Interventions: Other: MV Replacement
- MMR MV Repair: This group of patients had been randomized in the MMR study to mitral valve repair with annuloplasty ring.
  Interventions: Other: MV Repair
- CABG: This group of patients had been randomized in the MMR study to receive CABG
  Interventions: Other: CABG

INTERVENTIONS:
Other: MV Repair — Participants underwent mitral valve repair with annuloplasty and a sub-valvular procedure for severe tethering.
  Other Names: Mitral Valve Repair
  Groups: MMR MV Repair; SMR MV Repair
Other: MV Replacement — Participants underwent mitral valve replacement and complete preservation of the sub-valvular apparatus.
  Other Names: Mitral Valve Replacement
  Groups: MV Replacement
Other: CABG — Participants underwent coronary artery bypass grafting
  Other Names: Coronary Artery Bypass Grafting
  Groups: CABG

SUMMARY:
This study is a continuation of two previous studies --- the Severe Ischemic Mitral Regurgitation (SMR) Trial (NCT00807040) and the Moderate Ischemic Mitral regurgitation (MMR) Trial (NCT00806988) --- to learn more about patients' health 5-10 years after their mitral valve surgeries. The investigators will collect long-term health information on SMR and MMR trial participants using electronic medical records, patient and/or family input, public records, and healthcare- and vital status-related databases.

DETAILED DESCRIPTION:
This study is a continuation of two CTSN randomized trials --- the Severe Ischemic Mitral Regurgitation (SMR) Trial (NCT00807040) and the Moderate Ischemic Mitral regurgitation (MMR) Trial (NCT00806988) --- for the purpose of assessing the long-term outcomes of the index surgical therapies. Key clinical outcomes will be collected utilizing electronic medical records, patient and/or family input, public records, and healthcare- and vital status-related databases. Extended follow-up data will be obtained on up to 199 SMR and 270 MMR trial participants, who were alive at their 2-year follow-up evaluation. Patients will be followed for a minimum of 5 years and up to 10 years after randomization (the time of index surgical procedure). This follow-up data collection will be conducted by the Cardiothoracic Surgical Trials Network (CTSN) primarily utilizing the minimal PHI necessary to link data obtained from the MMR and SMR trials to other healthcare- and/or vital status-related databases.

Because the design of surgical trials for ischemic mitral regurgitation that would use mortality as a primary endpoint requires the enrollment of thousands of patients, the selected primary endpoint for the CTSN SMR and MMR trials was an echocardiographic measure of left ventricular remodeling. Secondary endpoints included, among others, survival, adverse events, readmissions and costs over a 2-year period. The SMR trial showed no difference in left ventricular reverse remodeling, but the rate of moderate or severe mitral regurgitation recurrence was significantly higher with mitral valve repair, resulting in more heart failure-related adverse events and cardiovascular admissions. Longer-term follow-up will be critical to assess whether this observed trend amongst SMR patients will continue and whether a survival difference will manifest over time. In moderate ischemic mitral regurgitation, mitral valve repair provided a more durable correction of mitral regurgitation than coronary artery bypass grafting (CABG) alone, but repair did not improve survival or reduce overall adverse events or readmissions, and was associated with an early hazard of neurological and supraventricular arrhythmic events. Longer-term follow-up of MMR patients will provide insights into whether the higher degree of recurrent mitral regurgitation with CABG alone will be associated with differences in adverse events, readmissions and survival. Additionally, the benefits of alternative surgical treatments for ischemic mitral regurgitation, which have differential upfront risks and costs, will likely extend beyond 2 years. Cost-effectiveness analysis will delineate the long-term cost-benefit trade-offs between mitral valve repair versus replacement for SMR, and of CABG with repair versus CABG alone for MMR, which should inform surgical decision making, and examine how differences in life expectancy and risk profiles of different patient groups affect cost-effectiveness over time. This extended follow-up should provide important clinical and health policy insights.

ELIGIBILITY:
Inclusion Criteria:

* Randomized patients in the MMR and SMR trials who were still alive at 2 years after the index cardiac surgical intervention

Exclusion Criteria:

* Patients participating in the MMR and SMR trials who withdrew consent prior to the 2-year follow-up evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Randomized patients in the MMR and SMR trials who were still alive at 2 years after the index cardiac surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Survival | up to 10 years post-surgery (at the time of registry data transfer)
  All-cause mortality will be assessed.

SECONDARY OUTCOMES:
Repeat Cardiac Interventions for MR | up to 10 years post-surgery (at the time of registry data transfer)
  Repeat cardiac interventions for MR in particular will be determined for the duration of follow-up and will be analyzed using a time-to-event analysis.
Hospital Costs | up to 10 years post-surgery (at the time of registry data transfer)
  Hospital costs will be calculated for the duration of follow-up utilizing the minimum PHI necessary to link the CTSN databases to other databases (e.g., Vizient, CMS Medicare, and Canadian Province databases). Cost data will be extracted from the Vizient operational database system for member sites or national payer or state-wide databases. Dates of charges and revenue codes will be used to match the cost data with data on readmissions. We will estimate costs including center-specific ratios of cost to charges. These ratios will be based on the annual Medicare costs reports submitted annually by participating study sites to Medicare. These data will be used to impute data for patients treated at hospitals, which are non-Vizient members.
Cost Effectiveness | up to 10 years post-surgery (at the time of registry data transfer)
  Cost Effectiveness using Incremental Cost Effectiveness Ratio and Net Health Benefit parameters. The primary objective of the cost-effectiveness analysis (CEA) is to estimate the incremental cost-effectiveness ratio (ICER) of the intervention under investigation as compared to the study-defined alternative. This ratio measures the ratio of the difference in costs and outcomes between the two study arms for each trial, with outcomes measured as life-years. We will also compute net health benefits (NHB) as an alternative way of looking at cost-effectiveness. This parameter compares the incremental effectiveness of an intervention with the minimum health effect that society would demand in return for the investment; i.e., with the health produced by investing at the societal ceiling cost-effectiveness ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Annetine C Gelijns, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Richard Weisel, MD, Study Chair — Toronto General Hospital
Locations (24):
- United States (16):
  - University of Southern California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Research Institute, Plano, Texas
  - University of Virginia Health Systems, Charlottesville, Virginia
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Canada (8):
  - University of Alberta Hospital, Edmonton, Alberta
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie de Quebec (Hopital Laval), Québec

IPD SHARING:
Plan to Share IPD: No